CLINICAL TRIAL: NCT07013435
Title: Thriving Beyond Treatment: A Resilience-Based Approach to Improve Long-term Quality of Life in Post-treatment Lymphoma Survivorship.
Brief Title: A Resilience-Based Approach to Improve Long-term Quality of Life in Post-treatment Lymphoma Survivorship
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Giselle K. Perez Lougee, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-204
Record Dates: First submitted 2025-05-23; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma
Keywords: quality of life; psychosocial intervention; supportive care; cancer survivorship; resilience
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education Program (Active Comparator): Participants will participate in 8 weekly sessions.
  Components include:
  * education on the co-occurrence of mental and physical problems
  * goal setting for health behavior change
  * self-monitoring
  HEP is an active control condition for mind body programs and is structurally equivalent to SMART3RP
  Interventions: Other: Health Education Program
- SMART3RP-Lymphoma (Experimental): Participants will participate in 8 weekly sessions.
  The intervention components include:
  * Eliciting the relaxation response (RR),
  * CBT strategies to improve stress management
  * Positive psychology strategies to achieve growth enhancement
  Interventions: Other: SMART3RP-Lymphoma

INTERVENTIONS:
Other: Health Education Program — 8 weekly sessions that include education on the co-occurrence of mental and physical problems, goal setting for health behavior change, and self-monitoring. Each session includes basic didactic information, interactive application of the information, and open discussion of didactic material.
  Arms: Health Education Program
Other: SMART3RP-Lymphoma — The SMART3RP-lymphoma is a group program that, through a variety of mind-body approaches, such as imagery, relaxation, and yoga, seeks to buffer stress and promote psychological resiliency and physical well-being.
  Arms: SMART3RP-Lymphoma

SUMMARY:
The goal of this trial is to learn if a resilience intervention can lead to improvements in lymphoma survivors' quality of life.

DETAILED DESCRIPTION:
The Stress Management and Relaxation Response Resiliency Program for lymphoma survivors (SMART3RP-Lymphoma) was adapted by researchers at the MGH. This group program seeks to buffer stress and promote psychological resiliency and physical well-being through a variety of mind-body approaches, such as imagery, relaxation, and yoga, cognitive behavioral strategies, and positive psychology tools.

The main questions it aims to answer are:

* Will survivors randomized to SMART3RP-Lymphoma demonstrate greater improvements in quality of life when compared to survivors randomized to a Health Education Program?
* Will improvements in resiliency lead to improvements in quality of life?

To answer these questions, researchers will compare a resilience intervention tailored to the needs of lymphoma survivors (SMART3RP-Lymphoma) to a Health Education Program to see how they affect quality of life of lymphoma survivors.

Participants will:

* Fill out 4 surveys across 12 months
* Participate in 8 weekly, virtual group sessions
* Submit hair cortisol samples

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking adults (18+ at time of enrollment)
* Within 2 years of completing active, curative treatment for lymphoma (includes surgery, chemotherapy, immunotherapy, radiation therapy, or other)

Exclusion Criteria:

* Active psychiatric or cognitive comorbidity as determined by the site PI or treating clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL): Change in PROMIS-29 | From enrollment to 6 month follow up
  To examine the effects of the SMART3RP-Lymphoma vs. a Health Education Program (HEP) in improving quality of life in early posttreatment lymphoma survivors. Quality of life will be measured using the PROMIS-29 which assesses physical, functional, emotional, and social quality of life. Each survey item is measured on a 1-5 scale. The unit of measurement is a score on a scale.

SECONDARY OUTCOMES:
Resilience: Change in Scores on the Current Experiences Scale (CES) | Enrollment to 3 month follow up
  To compare the effects of the SMART3RP-Lymphoma vs. a Health Education Program (HEP) on resilience in posttreatment lymphoma survivors. Resilience will be measured by the Current Experiences Scale (CES). The CES is a 23-item measure that assesses the following domains of resilience on 0-5 scale: appreciation for life, adaptive perspectives, personal strength, spiritual connectedness, relating to others, and health behaviors. The unit of measurement is a score on a scale.

OTHER OUTCOMES:
Correlation between scores on measures of Resilience (CES) and Quality of Life (PROMIS-29) | 3, 6 and 12 months
  We will determine how resilience at 3 months correlates to quality-of-life improvements at 6 and 12 months. Resilience will be measured by the Current Experiences Scale (CES), which is a 23-item measure. The CES assesses 6 domains of resilience including appreciation for life, adaptive perspectives, personal strength, spiritual connectedness, relating to others, and health behaviors). Quality of life will be measured by the PROMIS-29 which is a 29-item measure. It assesses physical, functional, emotional, and social quality of life domains. The unit of measurement for both assessments are scores on a scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified information as required by the NIH
Supporting Information: Study Protocol, SAP
Time Frame: Information will be made available as required by the NIH in public repository and via clinicaltrials.gov
Access Criteria: Researchers submitting formal requests as required and allowable by the NIH will be able to access supporting information.